CLINICAL TRIAL: NCT05737212
Title: A Multi-centered, Radiation Dose Escalation, Open, Exploratory, Phase 1/2a Clinical Trial on the Safety, Efficacy and Pharmacokinetic Characteristics of BNCT(Boron Neutron Capture Therapy) in Patients With Recurrent High-grade Gliomas
Brief Title: Studying the Safety, Efficacy, and Pharmacokinetic Characteristics of BNCT in Patients With Recurrent High-grade Gliomas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Phase 1 clinical trial was completed, and the study was stopped to initiate a Phase 2 trial with a revised protocol.
Sponsor: Dawonmedax Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM-BNCT-P001
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2023-02

CONDITIONS: Recurrent High-grade Glioma; Recurrent Glioblastoma; Recurrent Anaplastic Astrocytoma; Recurrent Anaplastic Oligodendroglioma
Keywords: Boron neutron capture therapy; boronophenylalanine; neutron capture therapy
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Oligodendroglioma

STUDY DESIGN:
Intervention Model Description: In the Phase I clinical study, the 3+3 dose escalation design is applied to evaluate the dose limiting toxicity (DLT) and 3 study subjects are enrolled to each group (Group 1, Group 2, Group 3). Depending on whether or not DLT occurs, 3 subjects at minimum to 18 subjects at maximum are enrolled.
  However, in the event a subject assigned a subject number withdraws from the study before starting BNCT or within 90 days from starting BNCT for reasons other than safety, up to 3 additional subjects can be enrolled for each dose group, resulting in 27 subjects at maximum allowed for enrollment for the Phase I clinical study.
  In the Phase IIa clinical study, up to 12 subjects are enrolled. However, subjects who are included in a group that has received the radiation dose confirmed as the maximum tolerated dose (MTD) in the Phase 1 clinical study AND satisfy all inclusion/exclusion criteria of the Phase IIa are included in the number of subjects of Phase IIa.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Radiation dose: 9 Gy-Eq
  * Investigational product, boronophenylalanine, DMX-101 500mg/kg/3hr
  * Investigational Device, DM-BTPS, DM-BNCT - neutron irradiation to reach maximum BNCT dose in brain of 9 Gy-Eq
  Interventions: Radiation: 500mg/kg/3hr followed by neutron irradiation to reach maximum brain dose of 9Gy-Eq
- Group 2 (Experimental): Radiation dose: 11 Gy-Eq
  * Investigational product, boronophenylalanine, DMX-101 500mg/kg/3hr
  * Investigational Device, DM-BTPS, DM-BNCT - neutron irradiation to reach maximum BNCT dose in brain of 11 Gy-Eq
  Interventions: Radiation: 500mg/kg/3hr followed by neutron irradiation to reach maximum brain dose of 11Gy-Eq
- Group 3 (Experimental): Radiation dose: 13 Gy-Eq
  * Investigational product, boronophenylalanine, DMX-101 500mg/kg/3hr
  * Investigational Device, DM-BTPS, DM-BNCT - neutron irradiation to reach maximum BNCT dose in brain of 13Gy-Eq
  Interventions: Radiation: 500mg/kg/3hr followed by neutron irradiation to reach maximum brain dose of 13Gy-Eq

INTERVENTIONS:
Radiation: 500mg/kg/3hr followed by neutron irradiation to reach maximum brain dose of 9Gy-Eq — Patients will be infused DMX-101 intravenously at a dose of 500mg/kg/hr over 3 hours. Thereafter, patient will receive neutron irradiation simultaneously for a certain period of time based on his Boronophenylalanine (BPA) concentration in the blood.
  Arms: Group 1
Radiation: 500mg/kg/3hr followed by neutron irradiation to reach maximum brain dose of 11Gy-Eq — Patients will be infused DMX-101 intravenously at a dose of 500mg/kg/hr over 3 hours. Thereafter, patient will receive neutron irradiation simultaneously for a certain period of time based on his Boronophenylalanine (BPA) concentration in the blood.
  Arms: Group 2
Radiation: 500mg/kg/3hr followed by neutron irradiation to reach maximum brain dose of 13Gy-Eq — Patients will be infused DMX-101 intravenously at a dose of 500mg/kg/hr over 3 hours. Thereafter, patient will receive neutron irradiation simultaneously for a certain period of time based on his Boronophenylalanine (BPA) concentration in the blood.
  Arms: Group 3

SUMMARY:
This is a multi-centered, radiation dose escalation, open, exploratory, Phase 1/2a clinical trial on the safety, efficacy and pharmacokinetic characteristics of BNCT in patients with recurrent high-grade gliomas.

The Phase I clinical study is to explore the adequate radiation dose level of BNCT based on confirmation of the maximum tolerated dose (radiation dose) of BNCT in patients with recurrent high-grade gliomas and characterize the safety, efficacy and pharmacokinetics.

To evaluate the primary objective of tolerability, subject population with history of exposure to a similar treatment recurrent high-grade glioma who received prior standard radiotherapy will be recruited.

The Phase IIa is to confirm the efficacy and safety after irradiation of radiation dose confirmed in the Phase I clinical study. To evaluate the primary objective of efficacy, subject population with glioblastoma (The 2021 WHO Classification of Tumors of the Central Nervous System, Glioblastoma IDH-wild type, WHO Grade 4) will be recruited.

DETAILED DESCRIPTION:
The subject receives the study drug administration and neutron irradiation in the BNCT clinic with all procedures performed under the control by the investigator affiliated to the study site. 500 mg/kg of the study drug is intravenously administered over 3 hours at a constant rate and neutron irradiation starts at 1 hour after the end of the study drug administration according to the previously established neutron irradiation plan.

All patients will be evaluated for response using magnetic resonance imaging (MRI) using RANO and modified RANO criteria.

ELIGIBILITY:
Inclusion Criteria:

1. An adult at the age 19 or above to under 80 at the time of written consent
2. Individual diagnosed with the following according to the WHO classification (2021)

   * Astrocytoma, IDH-mutant, WHO grade 3, 4
   * Oligodendroglioma, IDH-mutant, and 1p/19q-codeleted, WHO grade 3
   * Glioblastoma, IDH wildtype, WHO grade 4
   * Anaplastic Astrocytoma, NOS, WHO grade 3
   * Anaplastic Oligoastrocytoma, NOS, WHO grade 3
   * Anaplastic Oligodendroglioma, NOS, WHO grade 3
   * Glioblastoma, NOS, WHO grade 4
3. Individual who received radiation therapy at the standard level (54 to 66 Gy/25 to 35 fractions) or lower
4. Individual confirmed to have disease progression* according to the RANO criteria within 4 weeks from the screening visit (*) At least one lesion with contrast enhancement needs to exist on the contrast enhancement MRI. For a subject who shows no lesion with contrast enhancement, functional imaging such as 18F-FET or 18F-FDOPA PET/CT needs to confirm the existence of at least one clear recurrent lesion.

   However, in the event differentiation between recurrence and pseudoprogression is unclear, the subject cannot participate in the screening
5. Individual who is able to lie or sit for 30 minutes to 1 hour using the fixing device of the treatment couch
6. Individual with no metal implant such as a pacemaker
7. Individual with KPS (Karnofsky performance score) ≥ 60
8. Individual with an appropriate kidney function, lung function and bone marrow function based on the laboratory test at the screening visit

   * Hemoglobin ≥ 10.0 g/dL
   * WBC (white blood cell) ≥ 3,500/μL
   * Platelets ≥ 100,000/μL
   * Serum creatinine ≤ 1.5xULN
   * AST (aspartate aminotransferase)/ALT (alanine aminotransferase) ≤ 3xULN
9. Individual who receives sufficient explanation on the study, agrees to following the study procedures during the study period, and voluntarily decides to participate in the study and provides a written consent

   [Phase IIa study inclusion criteria]
10. Individual histologically diagnosed with glioblastoma
11. Individual with at least one measurable observed lesion according to the modified RANO criteria

Exclusion Criteria:

1. Individual to which a traditional therapy such as reoperation or reirradiation is effectively applicable based on consultation with a brain tumor multidisciplinary committee or consultation among two or more medical departments, including neurosurgery and radiation oncology
2. Individual who received cytotoxic anticancer therapy within 4 weeks from the screening visit (including previous interstitial anticancer therapy, local medication, and convection-enhanced delivery)
3. Individual who received targeted anticancer therapy (e.g., bevacizumab) within 6 weeks from the screening visit
4. Individual who received radiotherapy within 6 months from the screening visit
5. Individual who received a radical surgery for high-grade glioma within 4 weeks from the screening visit
6. Individual who received biopsy within 1 week from the screening visit
7. Individual confirmed to have a history of the following:

   * Interstitial brachytherapy
   * Stereotactic radiosurgery
   * Reirradiation for a recurrent lesion
   * Cancer immunotherapy
8. Individual with uncontrollable brain edema* even with the use of corticosteroid (*) Uncontrollable brain edema: Uncontrolled serious headache, vomiting, dyspnea, consciousness disturbance of NCI CTCAE (Ver. 5.0) grade 3 or above. However, for a patient taking corticosteroid, the patient must at least be on a stable dose or dose reduction for 7 days prior to the MRI scan at the screening visit.
9. Individual confirmed with meningeal dissemination
10. Individual diagnosed with cancer in another site* in the past at the time of the screening visit and whose disease-free period is less than 3 years (*) Patients with the skin basal cell carcinoma and carcinoma in situ of uterine cervix who received radical treatment are excluded
11. Individual with hypotonic dehydration or hereditary fructose intolerance
12. Individual with current or a history of phenylketonuria
13. Individual with serious infection (e.g., sepsis, HIV) in the opinion of the investigator
14. Individual who has dysfunction as below or, in the investigator's opinion, who is confirmed to have clinically significant disease (e.g., unstable angina, myocardial infarction) within 6 months from the screening visit:

    * Heart disease of Class II or above according to the New York Heart Association Functional Classification
    * Chronic obstructive pulmonary disease of moderate or higher severity according to the Chronic obstructive pulmonary disease clinical practice, or Dyspnea of Grade II or above according to the American thoracic society dyspnea scale
    * Hepatic dysfunction of Child-Pugh Classification B or C
15. Individual with current or a history of hypersensitivity to boron or any component of the study drug
16. Individual who received or applied other investigational product or device within 4 weeks from the screening visit
17. Individual who has received prior BNCT
18. Pregnant woman, breastfeeding woman, or individual who plans pregnancy or who does not agree to using and does not perform a medically reliable contraceptive method during the study period

    * Women of childbearing potential*: Use of 'intrauterine device', 'tubal surgery or tubal ligation', 'chemical barrier method (spermicide) + physical barrier method' or 'subcutaneously implanted contraceptive device + physical barrier method' (*) Woman of any potential of pregnancy, except for those who are before their first period, who received surgical sterilization (hysterectomy or bilateral ovariectomy) or who reached menopause (absence of menstrual periods for 12 months without any specific reason)
    * Male: Vasectomy or use of 'male condom + use of a medically reliable contraceptive method by the partner'
19. Individual not eligible for MRI or PET/CT scan
20. Individual the investigator otherwise considers ineligible for participating in the study [At the treatment planning visit, the following exclusion criteria will be checked:]
21. Individual not eligible for BNCT implementation according to the treatment plan established with DM-BTPS

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Phase I: To explore the adequate radiation dose level of BNCT based on confirmation of the maximum tolerated dose of BNCT | During 90 days post-BNCT
  To explore the adequate radiation dose level of BNCT based on confirmation of the maximum tolerated dose (radiation dose) of BNCT in patients with recurrent high-grade gliomas
Phase IIa: Proportion of 6-month PFS evaluated by central imaging according to the modified RANO criteria | 6 months
  Percentage of patients that are free from progressive disease for 6 months per modified RANO criteria

SECONDARY OUTCOMES:
Proportion of 6-month PFS evaluated by central imaging according to the RANO criteria | Up to 6 months
  Percentage of patients that are free from progressive disease for 6 months per RANO criteria
Proportion of 6-month PFS evaluated by the investigator according to the modified RANO criteria | Up to 6 months
  Percentage of patients that are free from progressive disease for 6 months per modified RANO criteria
Median PFS evaluated by central imaging according to the modified RANO criteria | Up to 6 months
  Median duration of progression free survival according to modified RANO criteria
Median PFS evaluated by central imaging according to the RANO criteria | Up to 6 months
  Median duration of progression free survival according to RANO criteria
Median PFS evaluated by the investigator according to the modified RANO criteria | Up to 6 months
  Median duration of progression free survival according to modified RANO criteria
ORR evaluated by central imaging according to the modified RANO criteria | Up to 6 months
  ORR will be defined as the percentage of patients with complete response (CR) or partial response (PR) according to the modified RANO criteria.
ORR evaluated by central imaging according to the RANO criteria | Up to 6 months
  ORR will be defined as the percentage of patients with complete response (CR) or partial response (PR) according to the RANO criteria.
ORR evaluated by the investigator according to the modified RANO criteria | Up to 6 months
  ORR will be defined as the percentage of patients with complete response (CR) or partial response (PR) according to the modified RANO criteria.
Median OS | Up to 2 years
  Median duration of overall survival for patients that are alive
Proportion of 1-year OS | Up to 2 years
  Percentage of patients that are alive for 1 year
Pharmacokinetic parameters(AUClast) of borono-phenylalanine in subjects with recurrent high-grade glioma | Based on whole blood sample up to 48 hours after the end of infusion
  The analysis is conducted using the Noncompartmental Analysis Method, and the results are summarized for each group in terms of descriptive statistics including the mean, standard deviation, minimum, median, and maximum values.
Pharmacokinetic parameters(AUCinf) of borono-phenylalanine in subjects with recurrent high-grade glioma | Based on whole blood sample up to 48 hours after the end of infusion
  The analysis is conducted using the Noncompartmental Analysis Method, and the results are summarized for each group in terms of descriptive statistics including the mean, standard deviation, minimum, median, and maximum values.
Pharmacokinetic parameters(Cmax) of borono-phenylalanine in subjects with recurrent high-grade glioma | Based on whole blood sample up to 48 hours after the end of infusion
  The analysis is conducted using the Noncompartmental Analysis Method, and the results are summarized for each group in terms of descriptive statistics including the mean, standard deviation, minimum, median, and maximum values.
Pharmacokinetic parameters(Tmax) of borono-phenylalanine in subjects with recurrent high-grade glioma | sampling up to 48 hours after the end of infusion
  The analysis is conducted using the Noncompartmental Analysis Method, and the results are summarized for each group in terms of descriptive statistics including the mean, standard deviation, minimum, median, and maximum values.
Pharmacokinetic parameters(CL) of borono-phenylalanine in subjects with recurrent high-grade glioma | Based on whole blood sample up to 48 hours after the end of infusion
  The analysis is conducted using the Noncompartmental Analysis Method, and the results are summarized for each group in terms of descriptive statistics including the mean, standard deviation, minimum, median, and maximum values.
Pharmacokinetic parameters(Vz) of borono-phenylalanine in subjects with recurrent high-grade glioma | Based on whole blood sample up to 48 hours after the end of infusion
  The analysis is conducted using the Noncompartmental Analysis Method, and the results are summarized for each group in terms of descriptive statistics including the mean, standard deviation, minimum, median, and maximum values.
Pharmacokinetic parameters(Vss) of borono-phenylalanine in subjects with recurrent high-grade glioma | Based on whole blood sample up to 48 hours after the end of infusion
  The analysis is conducted using the Noncompartmental Analysis Method, and the results are summarized for each group in terms of descriptive statistics including the mean, standard deviation, minimum, median, and maximum values.
Pharmacokinetic parameters(t1/2β) of borono-phenylalanine in subjects with recurrent high-grade glioma | Based on whole blood sample up to 48 hours after the end of infusion
  The analysis is conducted using the Noncompartmental Analysis Method, and the results are summarized for each group in terms of descriptive statistics including the mean, standard deviation, minimum, median, and maximum values.
Pharmacokinetic parameters(MRT) of borono-phenylalanine in subjects with recurrent high-grade glioma | Based on whole blood sample up to 48 hours after the end of infusion
  The analysis is conducted using the Noncompartmental Analysis Method, and the results are summarized for each group in terms of descriptive statistics including the mean, standard deviation, minimum, median, and maximum values.

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kim, M.D., Ph.D., Study Director — Dawonmedax Co., Ltd.
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No